CLINICAL TRIAL: NCT04489368
Title: Pathological Response Prediction to Neo-adjuvant Chemoradiotherapy in Esophageal Carcinoma and Comparison of Engineered Features Versus Deep Learning Models
Brief Title: Response Prediction to Neoadjuvant Chemoradiation in Esophageal Cancer Using Artificial Intelligence & Machine Learning
Acronym: QARC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dr Kundan Singh Chufal (Other)
Responsible Party: Sponsor-Investigator, Dr Kundan Singh Chufal, Senior Consultant & Chief of Thoracic Radiation Oncology, Department of Radiation Oncology, Rajiv Gandhi Cancer Institute & Research Center, India
Organization: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Other Study IDs: RGCIRC/IRB/80/2020
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Esophageal Neoplasm
Keywords: Artificial Intelligence; Deep Learning; Neoadjuvant Chemoradiation; Pathologic Response; Radiomics; Radiotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Esophagectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Patients undergoing NA-CCRT followed by Surgery
  Interventions: Radiation: Neo-Adjuvant Radiotherapy; Drug: Neo-Adjuvant Chemotherapy; Procedure: Esophagectomy

INTERVENTIONS:
Radiation: Neo-Adjuvant Radiotherapy — Neo-Adjuvant Radiotherapy via any technique, delivered concurrently with Neo-Adjuvant Chemotherapy.
Drug: Neo-Adjuvant Chemotherapy — Neo-Adjuvant Chemotherapy, delivered concurrently with Neo-Adjuvant Radiotherapy.
Procedure: Esophagectomy — Esophagectomy, performed 4-6 weeks after completion of Neo-Adjuvant Concurrent ChemoRadiation

SUMMARY:
In esophageal carcinoma, neoadjuvant concurrent chemo-radiotherapy (NA-CCRT) followed by surgery is the current standard of care and ample evidence has accumulated supporting the view that complete pathological response (pCR) is a positive prognostic marker for improved outcomes. Predicting the probability of achieving pCR prior to neoadjuvant treatment could permit modification of treatment protocols for those patients unlikely to achieve pCR.

Radiomics is a new entrant in the field of imaging where specific features are derived from the intensity and distribution pattern of pixels based on a region-of-interest (ROI). The features thus extracted can then be used for prediction modelling similar to other -omics datasets. Preliminary investigations examining its utility have been performed and its applications have thus far focused on screening and survival prediction after treatment. Due to the multi-dimensional nature of data extracted using radiomics, Artificial Intelligence (AI) methods are ideally suited for analysing and modelling radiomic features.

Machine Learning (ML) and Deep Learning (DL)[utilising Convolutional Neural Networks (CNN)] are both part of the AI framework. In contrast to ML, DL is a new entrant and has been utilised by some medical researchers for modelling using prediction-type algorithms. Besides significantly reducing the workflow associated with Radiomics-based research, feature engineering and modelling using DL are immune to the effects of incorrect ROI delineation. However, the main limitation of DL is the 'blackbox' effect, in which the underlying basis of a CNN is not known. This has been mitigated in part by the visualisation of activation maps directly on the image dataset to prove biological plausibility of predictions. The comparative performance of both types of modelling is also not known.

Our objective is to investigate pCR probability in our study population using radiomics-based ML and AI-based modelling. We will also investigate the comparative performance of both modelling techniques. For DL based prediction modelling, we will attempt to provide biological plausibility on the basis of activation maps.

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance Status: 0-2
* Patients with histopathological or cytopathological confirmed malignancy of the esophagus
* Histology: Squamous Cell Carcinoma and Adenocarcinoma
* Patients should have received NeoAdjuvant Concurrent Chemoradiation (NACCRT) followed by Surgery
* All therapeutic interventions (Radiotherapy, Chemotherapy & Surgery) delivered within participating institutions
* At least one pre-NACCRT DICOM imaging dataset (HRCT/ 18-FDG PET-CT/ Radiotherapy planning CT) for each patient

Exclusion Criteria:

* Patients with any metallic implants in the region of interest
* Patient with locally advanced disease or metastatic disease (T4 disease, Fistula, metastases)
* Patients with prior history of radiotherapy in the same region
* Patients developing a second malignancy in the esophagus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient records in each participating research center from January 2011 to 1st May 2020
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-01-16 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Develop models to predict pCR based on pre-neoadjuvant imaging modalities | August 2021
Perform a clinical audit of patient outcomes (OS, RFS, pCR rate) after new-adjuvant chemoradiation and esophagectomy | January 2020

CONTACTS AND LOCATIONS:
Overall Officials: Kundan S Chufal, MD, Principal Investigator — Rajiv Gandhi Cancer Institute & Research Center
Locations (2):
- Illawarra Cancer Care Centre, Wollongong, Australia
- Rajiv Gandhi Cancer Institute & Research Center, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No